CLINICAL TRIAL: NCT00196937
Title: Phase 3, Open, Age-stratified Study to Assess Immunogenicity and Safety of GSK Biologicals' HPV-16/18 Vaccine Administered Intramuscularly According to 3-dose Schedule (0,1,6 Months) in Healthy Female Subjects Aged 15 - 55 Years and Long Term Follow-up
Brief Title: Human Papilloma Virus (HPV) Vaccine Immunogenicity and Safety Trial in Young and Adult Women With GSK Biologicals' HPV-16/18
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 103514; 105879 (Other: GSK); 105880 (Other: GSK); 105881 (Other: GSK); 105882 (Other: GSK); 2004-002083-18 (EudraCT Number); NCT00332358 (obsolete NCT alias); NCT00332475 (obsolete NCT alias); NCT00332501 (obsolete NCT alias); NCT00332527 (obsolete NCT alias)
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Results first posted 2010-08-06 (Estimated); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Infections, Papillomavirus
Keywords: HPV Vaccine Safety
MeSH Terms: conditions — Papillomavirus Infections | interventions — human papillomavirus vaccine, L1 type 16, 18

ARMS (3):
- Cervarix (15-25 Years) Group (Experimental): Women aged 15 to 25 years received 3 doses of Cervarix vaccine administered according to a 0, 1, 6-month schedule.
  Interventions: Biological: Cervarix
- Cervarix (26-45 Years) Group (Experimental): Women aged 26 to 45 years received 3 doses of Cervarix vaccine administered according to a 0, 1, 6-month schedule.
  Interventions: Biological: Cervarix
- Cervarix (46-55 Years) Group (Experimental): Women aged 46 to 55 years received 3 doses of Cervarix vaccine administered according to a 0, 1, 6-month schedule.
  Interventions: Biological: Cervarix

INTERVENTIONS:
Biological: Cervarix — Three doses of vaccine administered intramuscularly according to a 0, 1, 6-month schedule.

SUMMARY:
Infection with human papillomavirus (HPV) has been clearly established as the central cause of cervical cancer. Indeed, certain oncogenic types of HPV can infect the cervix (part of the uterus or womb). This infection may go away by itself, but if it does not go away (this is called persistent infection), it can lead in women over a long period of time to cancer of the cervix. This study will evaluate the immunogenicity and safety of GSK Biologicals HPV-16/18 vaccine over 12 months, in women up to 55 years of age at study start. Approximately 660 study subjects will receive the HPV vaccine administered intramuscularly according to a 0-1-6 month schedule. The study will be extended to assess long-term safety and immunogenicity of the HPV-16/18 vaccine.

ELIGIBILITY:
Inclusion criteria for primary study:

* A woman who the investigator believes that she and/or her parents/legally acceptable representative can and will comply with the requirements of the protocol.
* A woman between, and including, 15 and 55 years of age at the time of the first vaccination.
* Written informed consent obtained from the subject prior to enrolment (for subjects below the legal age of consent, written informed consent must be obtained from a parent or legally acceptable representative and, in addition, the subject should sign and personally date a written informed assent).
* Free of obvious health problems.
* Subject must have a negative urine pregnancy test.
* Subject must be of non-childbearing potential or, if of childbearing potential, she must be abstinent or must be using adequate contraceptive precautions for 30 days prior to vaccination and must agree to continue such precautions for two months after completion of the vaccination series. Subjects who reach menarche during the study and therefore become of childbearing potential must agree to follow the same precautions

Inclusion criteria for extension studies

* A female who enrolled in the primary study and received three doses of vaccine.
* Written informed consent obtained from the subject prior to enrolment (for subjects below the legal age of consent, written informed consent must be obtained from a parent or legally acceptable representative and, in addition, the subject must sign and personally date a written informed assent).

Exclusion criteria for primary study:

* Pregnant or breastfeeding.
* A woman planning to become pregnant, likely to become pregnant (as determined by the investigator) or planning to discontinue contraceptive precautions during the study period, up to two months after the last vaccine dose.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period (up to Month 12).
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose, or planned administration during the study period.
* Planned administration/administration of a vaccine not foreseen by the study protocol within 30 days before and 30 days after the first dose of study vaccine. Planned administration/administration of routine vaccines up to 8 days before the first dose of study vaccine is allowed. Enrolment will be deferred until the subject is outside of specified window.
* Previous administration of components of the investigational vaccine
* Previous vaccination against HPV.
* Any medically diagnosed or suspected immunodeficient condition based on medical history and physical examination.
* History of allergic disease, suspected allergy or reactions likely to be exacerbated by any component of the study vaccine.
* Hypersensitivity to latex.
* Known acute or chronic, clinically significant neurologic, hepatic or renal functional abnormality, as determined by previous physical examination or laboratory tests.
* History of chronic condition(s) requiring treatment.
* Administration of immunoglobulins and/or any blood product within 3 months preceding the first dose of study vaccine or planned administration during the study period. Enrolment will be deferred until the subject is outside of specified window.
* Acute disease at the time of enrolment.

Exclusion criteria for extension studies

* Use of any investigational or non-registered product (drug or vaccine) or planned use during the study period.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* Chronic administration of immunosuppressants or other immune-modifying drugs occurring less than 3 months prior to blood sampling.
* Administration of immunoglobulins and/or any blood products within the three months preceding blood sampling.

Ages: 15 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 667 (Actual)
Dates: Start 2004-10-07 (Actual); Primary Completion 2005-12-15 (Actual); Study Completion 2005-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- Germany (3):
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Berlin
- Poland (2):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Poznan

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/Posting.aspx?ID=1513

REFERENCES:
- [Background] Descamps D, Hardt K, Spiessens B, Izurieta P, Verstraeten T, Breuer T, Dubin G. Safety of human papillomavirus (HPV)-16/18 AS04-adjuvanted vaccine for cervical cancer prevention: a pooled analysis of 11 clinical trials. Hum Vaccin. 2009 May;5(5):332-40. doi: 10.4161/hv.5.5.7211. Epub 2009 May 20. PMID 19221517
- [Background] Schwarz TF, Spaczynski M, Schneider A, Wysocki J, Galaj A, Perona P, Poncelet S, Zahaf T, Hardt K, Descamps D, Dubin G; HPV Study Group for Adult Women. Immunogenicity and tolerability of an HPV-16/18 AS04-adjuvanted prophylactic cervical cancer vaccine in women aged 15-55 years. Vaccine. 2009 Jan 22;27(4):581-7. doi: 10.1016/j.vaccine.2008.10.088. Epub 2008 Nov 18. PMID 19022320
- [Background] Schwarz TF, Spaczynski M, Schneider A, Wysocki J, Galaj A, Schulze K, Poncelet SM, Catteau G, Thomas F, Descamps D. Persistence of immune response to HPV-16/18 AS04-adjuvanted cervical cancer vaccine in women aged 15-55 years. Hum Vaccin. 2011 Sep;7(9):958-65. doi: 10.4161/hv.7.9.15999. Epub 2011 Sep 1. PMID 21892005
- [Background] Schwarz TF, Kocken M, Petaja T, Einstein MH, Spaczynski M, Louwers JA, Pedersen C, Levin M, Zahaf T, Poncelet S, Hardt K, Descamps D, Dubin G. Correlation between levels of human papillomavirus (HPV)-16 and 18 antibodies in serum and cervicovaginal secretions in girls and women vaccinated with the HPV-16/18 AS04-adjuvanted vaccine. Hum Vaccin. 2010 Dec;6(12):1054-61. doi: 10.4161/hv.6.12.13399. Epub 2010 Dec 1. PMID 21157180
- [Derived] Schwarz T, Spaczynski M, Kaufmann A, Wysocki J, Galaj A, Schulze K, Suryakiran P, Thomas F, Descamps D. Persistence of immune responses to the HPV-16/18 AS04-adjuvanted vaccine in women aged 15-55 years and first-time modelling of antibody responses in mature women: results from an open-label 6-year follow-up study. BJOG. 2015 Jan;122(1):107-18. doi: 10.1111/1471-0528.13070. Epub 2014 Sep 11. PMID 25208608
- [Derived] Boxus M, Lockman L, Fochesato M, Lorin C, Thomas F, Giannini SL. Antibody avidity measurements in recipients of Cervarix vaccine following a two-dose schedule or a three-dose schedule. Vaccine. 2014 May 30;32(26):3232-6. doi: 10.1016/j.vaccine.2014.04.005. Epub 2014 Apr 13. PMID 24731816
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 103514 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 103514 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register. The results of this study 103514 are summarised with studies 105880 and 105881 on the GSK Clinical Study Register.
- Available data/document: Clinical Study Report: 103514 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 103514 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 103514 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 103514 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 103514 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of the 667 enrolled subjects, 1 subject was excluded for not receiving vaccination and the actual starting number was 666.
Period: Overall Study
Arm/Group | Cervarix (15-25 Years) Group | Cervarix (26-45 Years) Group | Cervarix (46-55 Years) Group
Started | 229 | 226 | 211
Completed | 220 | 221 | 204
Not Completed | 9 | 5 | 7
Not completed — Serious Adverse Event | 1 | 0 | 0
Not completed — Non-serious adverse event | 1 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 2
Not completed — Lost to Follow-up | 4 | 3 | 3
Not completed — Other | 3 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cervarix (15-25 Years) Group | Cervarix (26-45 Years) Group | Cervarix (46-55 Years) Group | Total
Number analyzed (Participants) | 229 | 226 | 211 | 666
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.9 (2.67) | 35.5 (6.02) | 49.6 (2.80) | 34.9 (12.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 229 | 226 | 211 | 666
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 229 | 225 | 211 | 665
  Black | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroconverted Subjects for Anti-human Papilloma Virus 16 (Anti-HPV-16) and Anti-human Papilloma Virus 18 (Anti-HPV-18) Antibodies, in Women 15 to 25 Years of Age and Women 26 to 45 Years of Age
Description: Seroconversion was defined as the appearance of anti-HPV-16 and/or anti-HPV-18 antibodies [i.e. antibody titer greater than or equal to (≥) the cut-off value] in the sera of subjects seronegative before vaccination. Cut-off values were 8 enzyme-linked immunosorbent assay (ELISA) units per milliliter (EL.U/mL) for anti-HPV-16 antibodies and 7 EL.U/mL for anti-HPV-18 antibodies. Data for the Cervarix (46-55 Years) Group are presented in the Secondary Outcomes as per Protocol.
Time Frame: At Month 7
Population: The analysis was based the According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom immunogenicity data were available at the time of the analysis and who were seronegative before vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix (15-25 Years) Group | Cervarix (26-45 Years) Group
Number analyzed (Participants) | 202 | 185
Participants
  Anti-HPV-16: number analyzed (Participants) | 191 | 164
  Anti-HPV-16 | 191 | 164
  Anti-HPV-18 | 202 | 185
Statistical Analysis 1: Comparison: Cervarix (15-25 Years) Group vs Cervarix (26-45 Years) Group; Immune response to anti-HPV-16 in terms of SCR: To evaluate if the immunogenicity (as determined by ELISA) of the Cervarix vaccine, one month after the third dose (Month 7), in young women 26 - 45 years of age is non-inferior to that in women 15 - 25 years of age; Test type: Non-Inferiority — Non-inferiority with respect to seroconversion was shown if, for both anti-HPV-16 and anti-HPV-18 antibodies, the upper limit of the 95% confidence interval (CI) for the difference [Cervarix (15-25 years) Group minus Cervarix (26-45 years) Group] was below 10%; Difference in SCR = 0, 95% CI 2-sided [-1.97 to 2.29]
Statistical Analysis 2: Comparison: Cervarix (15-25 Years) Group vs Cervarix (26-45 Years) Group; Immune response to anti-HPV-18 in terms of SCR: To evaluate if the immunogenicity (as determined by ELISA) of the Cervarix vaccine, one month after the third dose (Month 7), in young women 26 - 45 years of age is non-inferior to that in women 15 - 25 years of age; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Difference in SCR = 0, 95% CI 2-sided [-1.87 to 2.03]

2. Primary Outcome: Anti-HPV-16/18 Antibody Titers Assessed by ELISA Based on the ATP Cohort for Immunogenicity at Months 18, 24, 36 and 48
Description: Anti-HPV 16/18 antibody titers were detected in sera samples and presented as Geometric Mean Titers (GMT), expressed in EL.U/mL. Data for pre-vaccination, Month 2, Month 7 and Month 12 are presented in the Secondary Outcomes as per Protocol.
Time Frame: At Months 18, 24, 36 and 48
Population: The analysis was based on the ATP cohort for immunogenicity, which included all evaluable subjects for whom immunogenicity data were available at the time of the analysis and who were seronegative before vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix (15-25 Years) Group | Cervarix (26-45 Years) Group | Cervarix (46-55 Years) Group
Number analyzed (Participants) | 224 | 219 | 201
EL.U/mL
  Anti-HPV-16 (Month 18): number analyzed (Participants) | 149 | 132 | 123
  Anti-HPV-16 (Month 18) | 2197.9 [1870.5 to 2582.6] | 933.3 [771.4 to 1129.1] | 578.5 [486.2 to 688.2]
  Anti-HPV-16 (Month 24): number analyzed (Participants) | 148 | 136 | 125
  Anti-HPV-16 (Month 24) | 1730.7 [1462.3 to 2048.5] | 733.0 [603.7 to 890.1] | 472.9 [396.8 to 563.6]
  Anti-HPV-16 (Month 36): number analyzed (Participants) | 141 | 129 | 118
  Anti-HPV-16 (Month 36) | 1491.5 [1260.9 to 1764.1] | 607.2 [502.8 to 733.3] | 363.9 [301.6 to 439.1]
  Anti-HPV-16 (Month 48): number analyzed (Participants) | 148 | 142 | 127
  Anti-HPV-16 (Month 48) | 1382.7 [1166.6 to 1638.9] | 524.2 [437.7 to 627.9] | 324.0 [272.2 to 385.5]
  Anti-HPV-18 (Month 18): number analyzed (Participants) | 156 | 146 | 156
  Anti-HPV-18 (Month 18) | 816.0 [694.1 to 959.3] | 328.4 [275.3 to 391.7] | 247.9 [210.1 to 292.4]
  Anti-HPV-18 (Month 24): number analyzed (Participants) | 151 | 153 | 156
  Anti-HPV-18 (Month 24) | 673.6 [568.3 to 798.4] | 280.8 [235.3 to 335.1] | 185.7 [156.3 to 220.6]
  Anti-HPV-18 (Month 36): number analyzed (Participants) | 14 | 148 | 150
  Anti-HPV-18 (Month 36) | 539.9 [280.6 to 1038.8] | 220.1 [184.5 to 262.5] | 136.9 [114.9 to 163.0]
  Anti-HPV-18 (Month 48): number analyzed (Participants) | 154 | 156 | 156
  Anti-HPV-18 (Month 48) | 475.5 [400.9 to 564.1] | 189.0 [159.3 to 224.2] | 122.9 [102.3 to 147.6]

3. Secondary Outcome: Number of Seroconverted Subjects for Anti-HPV-16 and Anti-HPV-18 Antibodies, in Women 46 - 55 Years of Age
Description: Seroconversion was defined as the appearance of anti-HPV-16 and/or anti-HPV-18 antibodies (i.e. antibody titer ≥ cut-off value) in the sera of subjects seronegative before vaccination. Cut-off values were 8 EL.U/mL for anti-HPV-16 antibodies and 7 EL.U/mL for anti-HPV-18 antibodies. Seroconversion results at Month 7 for the Cervarix (15-25 Years) Group and for the Cervarix (26-45 Years) Group are presented in the Primary Outcome Measure 1.
Time Frame: At Month 7
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix (46-55 Years) Group
Number analyzed (Participants) | 172
Participants
  Anti-HPV-16: number analyzed (Participants) | 136
  Anti-HPV-16 | 136
  Anti-HPV-18 | 172

4. Secondary Outcome: Anti-HPV-16/18 Antibody Titers Assessed by ELISA Based on the ATP Cohort for Immunogenicity at Pre-vaccination (PRE) and Months 2, 7 and 12
Description: Anti-HPV 16/18 antibody titers were detected in sera samples and presented as GMT, expressed in EL.U/mL. Data for Months 18, 24, 36 and 48 are presented in the Primary Outcome Measure 2 as per Protocol.
Time Frame: At PRE and Months 2, 7 and 12
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix (15-25 Years) Group | Cervarix (26-45 Years) Group | Cervarix (46-55 Years) Group
Number analyzed (Participants) | 224 | 219 | 201
EL.U/mL
  Anti-HPV-16 (PRE): number analyzed (Participants) | 195 | 164 | 139
  Anti-HPV-16 (PRE) | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0]
  Anti-HPV-16 (Month 2): number analyzed (Participants) | 195 | 164 | 139
  Anti-HPV-16 (Month 2) | 3090.0 [2791.9 to 3419.9] | 1824.6 [1600.5 to 2080.1] | 1269.9 [1100.1 to 1465.9]
  Anti-HPV-16 (Month 7): number analyzed (Participants) | 191 | 164 | 136
  Anti-HPV-16 (Month 7) | 7908.4 [6874.0 to 9098.5] | 4029.2 [3402.7 to 4771.0] | 2566.8 [2181.2 to 3020.6]
  Anti-HPV-16 (Month 12): number analyzed (Participants) | 183 | 163 | 134
  Anti-HPV-16 (Month 12) | 3055.3 [2620.4 to 3562.4] | 1563.7 [1313.4 to 1861.8] | 926.2 [787.2 to 1089.7]
  Anti-HPV-18 (PRE): number analyzed (Participants) | 207 | 186 | 175
  Anti-HPV-18 (PRE) | 3.5 [3.5 to 3.5] | 3.5 [3.5 to 3.5] | 3.5 [3.5 to 3.5]
  Anti-HPV-18 (Month 2): number analyzed (Participants) | 207 | 186 | 175
  Anti-HPV-18 (Month 2) | 2229.0 [1995.0 to 2490.5] | 1390.3 [1230.2 to 1571.2] | 957.2 [842.2 to 1088.0]
  Anti-HPV-18 (Month 7): number analyzed (Participants) | 202 | 185 | 172
  Anti-HPV-18 (Month 7) | 3499.3 [3098.7 to 3951.6] | 1837.3 [1602.1 to 2107.0] | 1313.0 [1145.6 to 1504.9]
  Anti-HPV-18 (Month 12): number analyzed (Participants) | 192 | 182 | 169
  Anti-HPV-18 (Month 12) | 1284.6 [1112.7 to 1483.2] | 619.8 [526.8 to 729.2] | 430.2 [370.5 to 499.7]

5. Secondary Outcome: Number of Subjects Seroconverted for Anti-HPV-16 and Anti-HPV-18 Antibodies at Month 2 and Month 12
Description: Seroconversion was defined as the appearance of anti-HPV-16 and/or anti- HPV-18 antibodies (i.e. antibody titer ≥ cut-off value) in the sera of subjects seronegative before vaccination. Cut-off values were 8 EL.U/mL for anti-HPV-16 antibodies and 7 EL.U/mL for anti-HPV-18 antibodies. Seroconversion results at Month 7 are presented in the Primary Outcome Measure 1 for Cervarix (15-25 Years) Group and Cervarix (26-45 Years) Group and in the Secondary Outcome Measure 3 for the Cervarix (46-55 Years) Group.
Time Frame: At Month 2 and Month 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix (15-25 Years) Group | Cervarix (26-45 Years) Group | Cervarix (46-55 Years) Group
Number analyzed (Participants) | 207 | 186 | 175
Participants
  Anti-HPV-16 (Month 2): number analyzed (Participants) | 195 | 164 | 139
  Anti-HPV-16 (Month 2) | 195 | 164 | 139
  Anti-HPV-16 (Month 12): number analyzed (Participants) | 183 | 163 | 134
  Anti-HPV-16 (Month 12) | 183 | 163 | 134
  Anti-HPV-18 (Month 2) | 207 | 186 | 175
  Anti-HPV-18 (Month 12): number analyzed (Participants) | 192 | 182 | 169
  Anti-HPV-18 (Month 12) | 192 | 182 | 169

6. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were arthralgia, fatigue, fever, gastrointestinal symptoms, headache, myalgia, rash and urticaria. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever above (>) 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 7-day period (from the day of vaccination up to 6 subsequent days) following vaccination after each dose and across doses
Population: The analysis was based on the Total Vaccinated Cohort (TVC), which included all subjects with at least one study vaccine administered, on subjects with symptom sheets completed and for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix (15-25 Years) Group | Cervarix (26-45 Years) Group | Cervarix (46-55 Years) Group
Number analyzed (Participants) | 227 | 226 | 207
Participants
  Any Arthralgia - Dose 1: number analyzed (Participants) | 226 | 226 | 207
  Any Arthralgia - Dose 1 | 21 | 15 | 22
  Any Arthralgia - Dose 2: number analyzed (Participants) | 227 | 224 | 207
  Any Arthralgia - Dose 2 | 17 | 22 | 26
  Any Arthralgia - Dose 3: number analyzed (Participants) | 217 | 218 | 199
  Any Arthralgia - Dose 3 | 22 | 20 | 22
  Any Arthralgia - Across doses | 45 | 43 | 47
  Grade 3 Arthralgia - Dose 1: number analyzed (Participants) | 226 | 226 | 207
  Grade 3 Arthralgia - Dose 1 | 0 | 0 | 1
  Grade 3 Arthralgia - Dose 2: number analyzed (Participants) | 227 | 224 | 207
  Grade 3 Arthralgia - Dose 2 | 1 | 3 | 0
  Grade 3 Arthralgia - Dose 3: number analyzed (Participants) | 217 | 218 | 199
  Grade 3 Arthralgia - Dose 3 | 0 | 0 | 1
  Grade 3 Arthralgia - Across doses | 1 | 3 | 2
  Related Arthralgia - Dose 1: number analyzed (Participants) | 226 | 226 | 207
  Related Arthralgia - Dose 1 | 14 | 7 | 9
  Related Arthralgia - Dose 2: number analyzed (Participants) | 227 | 224 | 207
  Related Arthralgia - Dose 2 | 11 | 9 | 12
  Related Arthralgia - Dose 3: number analyzed (Participants) | 217 | 218 | 199
  Related Arthralgia - Dose 3 | 14 | 11 | 8
  Related Arthralgia - Across doses | 28 | 23 | 22
  Any Fatigue - Dose 1: number analyzed (Participants) | 226 | 226 | 207
  Any Fatigue - Dose 1 | 85 | 72 | 47
  Any Fatigue - Dose 2: number analyzed (Participants) | 227 | 224 | 207
  Any Fatigue - Dose 2 | 68 | 53 | 48
  Any Fatigue - Dose 3: number analyzed (Participants) | 217 | 218 | 199
  Any Fatigue - Dose 3 | 84 | 68 | 50
  Any Fatigue - Across doses | 128 | 116 | 81
  Grade 3 Fatigue - Dose 1: number analyzed (Participants) | 226 | 226 | 207
  Grade 3 Fatigue - Dose 1 | 0 | 2 | 1
  Grade 3 Fatigue - Dose 2: number analyzed (Participants) | 227 | 224 | 207
  Grade 3 Fatigue - Dose 2 | 3 | 0 | 2
  Grade 3 Fatigue - Dose 3: number analyzed (Participants) | 217 | 218 | 199
  Grade 3 Fatigue - Dose 3 | 2 | 0 | 1
  Grade 3 Fatigue - Across doses | 5 | 2 | 4
  Related Fatigue - Dose 1: number analyzed (Participants) | 226 | 226 | 207
  Related Fatigue - Dose 1 | 46 | 34 | 25
  Related Fatigue - Dose 2: number analyzed (Participants) | 227 | 224 | 207
  Related Fatigue - Dose 2 | 46 | 24 | 23
  Related Fatigue - Dose 3: number analyzed (Participants) | 217 | 218 | 199
  Related Fatigue - Dose 3 | 54 | 40 | 30
  Related Fatigue - Across doses | 86 | 60 | 44
  Any Fever - Dose 1: number analyzed (Participants) | 226 | 226 | 207
  Any Fever - Dose 1 | 10 | 7 | 2
  Any Fever - Dose 2: number analyzed (Participants) | 227 | 224 | 207
  Any Fever - Dose 2 | 9 | 7 | 2
  Any Fever - Dose 3: number analyzed (Participants) | 217 | 218 | 199
  Any Fever - Dose 3 | 5 | 8 | 2
  Any Fever - Across doses | 128 | 116 | 81
  Grade 3 Fever - Dose 1: number analyzed (Participants) | 226 | 226 | 207
  Grade 3 Fever - Dose 1 | 0 | 1 | 0
  Grade 3 Fever - Dose 2: number analyzed (Participants) | 227 | 224 | 207
  Grade 3 Fever - Dose 2 | 0 | 0 | 0
  Grade 3 Fever - Dose 3: number analyzed (Participants) | 217 | 218 | 199
  Grade 3 Fever - Dose 3 | 0 | 0 | 0
  Grade 3 Fever - Across doses | 0 | 1 | 0
  Related Fever - Dose 1: number analyzed (Participants) | 226 | 226 | 207
  Related Fever - Dose 1 | 7 | 3 | 1
  Related Fever - Dose 2: number analyzed (Participants) | 227 | 224 | 207
  Related Fever - Dose 2 | 4 | 1 | 1
  Related Fever - Dose 3: number analyzed (Participants) | 217 | 218 | 199
  Related Fever - Dose 3 | 2 | 2 | 1
  Related Fever - Across doses | 11 | 6 | 3
  Any Gastrointestinal - Dose 1: number analyzed (Participants) | 226 | 226 | 207
  Any Gastrointestinal - Dose 1 | 34 | 18 | 12
  Any Gastrointestinal - Dose 2: number analyzed (Participants) | 227 | 224 | 207
  Any Gastrointestinal - Dose 2 | 25 | 11 | 14
  Any Gastrointestinal - Dose 3: number analyzed (Participants) | 217 | 218 | 199
  Any Gastrointestinal - Dose 3 | 16 | 14 | 12
  Any Gastrointestinal - Across doses | 51 | 33 | 31
  Grade 3 Gastrointestinal - Dose 1: number analyzed (Participants) | 226 | 226 | 207
  Grade 3 Gastrointestinal - Dose 1 | 1 | 3 | 1
  Grade 3 Gastrointestinal - Dose 2: number analyzed (Participants) | 227 | 224 | 207
  Grade 3 Gastrointestinal - Dose 2 | 0 | 0 | 0
  Grade 3 Gastrointestinal - Dose 3: number analyzed (Participants) | 217 | 218 | 199
  Grade 3 Gastrointestinal - Dose 3 | 0 | 0 | 2
  Grade 3 Gastrointestinal - Across doses | 1 | 3 | 3
  Related Gastrointestinal - Dose 1: number analyzed (Participants) | 226 | 226 | 207
  Related Gastrointestinal - Dose 1 | 22 | 4 | 7
  Related Gastrointestinal - Dose 2: number analyzed (Participants) | 227 | 224 | 207
  Related Gastrointestinal - Dose 2 | 15 | 6 | 6
  Related Gastrointestinal - Dose 3: number analyzed (Participants) | 217 | 218 | 199
  Related Gastrointestinal - Dose 3 | 11 | 10 | 5
  Related Gastrointestinal - Across doses | 30 | 15 | 16
  Any Headache - Dose 1: number analyzed (Participants) | 226 | 226 | 207
  Any Headache - Dose 1 | 77 | 62 | 50
  Any Headache - Dose 2: number analyzed (Participants) | 227 | 224 | 207
  Any Headache - Dose 2 | 63 | 43 | 44
  Any Headache - Dose 3: number analyzed (Participants) | 217 | 218 | 199
  Any Headache - Dose 3 | 64 | 47 | 39
  Any Headache - Across doses | 123 | 100 | 82
  Grade 3 Headache - Dose 1: number analyzed (Participants) | 226 | 226 | 207
  Grade 3 Headache - Dose 1 | 3 | 3 | 0
  Grade 3 Headache - Dose 2: number analyzed (Participants) | 227 | 224 | 207
  Grade 3 Headache - Dose 2 | 5 | 3 | 2
  Grade 3 Headache - Dose 3: number analyzed (Participants) | 217 | 218 | 199
  Grade 3 Headache - Dose 3 | 4 | 1 | 4
  Grade 3 Headache - Across doses | 10 | 5 | 6
  Related Headache - Dose 1: number analyzed (Participants) | 226 | 226 | 207
  Related Headache - Dose 1 | 42 | 27 | 25
  Related Headache - Dose 2: number analyzed (Participants) | 227 | 224 | 207
  Related Headache - Dose 2 | 34 | 25 | 17
  Related Headache - Dose 3: number analyzed (Participants) | 217 | 218 | 199
  Related Headache - Dose 3 | 40 | 25 | 23
  Related Headache - Across doses | 77 | 48 | 46
  Any Myalgia - Dose 1: number analyzed (Participants) | 226 | 226 | 207
  Any Myalgia - Dose 1 | 93 | 49 | 48
  Any Myalgia - Dose 2: number analyzed (Participants) | 227 | 224 | 207
  Any Myalgia - Dose 2 | 69 | 50 | 42
  Any Myalgia - Dose 3: number analyzed (Participants) | 217 | 218 | 199
  Any Myalgia - Dose 3 | 71 | 64 | 41
  Any Myalgia - Across doses | 126 | 97 | 83
  Grade 3 Myalgia - Dose 1: number analyzed (Participants) | 226 | 226 | 207
  Grade 3 Myalgia - Dose 1 | 1 | 0 | 2
  Grade 3 Myalgia - Dose 2: number analyzed (Participants) | 227 | 224 | 207
  Grade 3 Myalgia - Dose 2 | 4 | 5 | 1
  Grade 3 Myalgia - Dose 3: number analyzed (Participants) | 217 | 218 | 199
  Grade 3 Myalgia - Dose 3 | 4 | 6 | 1
  Grade 3 Myalgia - Across doses | 8 | 9 | 4
  Related Myalgia - Dose 1: number analyzed (Participants) | 226 | 226 | 207
  Related Myalgia - Dose 1 | 71 | 32 | 30
  Related Myalgia - Dose 2: number analyzed (Participants) | 227 | 224 | 207
  Related Myalgia - Dose 2 | 52 | 28 | 23
  Related Myalgia - Dose 3: number analyzed (Participants) | 217 | 218 | 199
  Related Myalgia - Dose 3 | 58 | 38 | 20
  Related Myalgia - Across doses | 96 | 62 | 48
  Any Rash - Dose 1: number analyzed (Participants) | 226 | 226 | 207
  Any Rash - Dose 1 | 6 | 7 | 4
  Any Rash - Dose 2: number analyzed (Participants) | 227 | 224 | 207
  Any Rash - Dose 2 | 4 | 4 | 3
  Any Rash - Dose 3: number analyzed (Participants) | 217 | 218 | 199
  Any Rash - Dose 3 | 10 | 5 | 1
  Any Rash - Across doses | 16 | 14 | 7
  Grade 3 Rash - Dose 1: number analyzed (Participants) | 226 | 226 | 207
  Grade 3 Rash - Dose 1 | 0 | 0 | 0
  Grade 3 Rash - Dose 2: number analyzed (Participants) | 227 | 224 | 207
  Grade 3 Rash - Dose 2 | 0 | 0 | 0
  Grade 3 Rash - Dose 3: number analyzed (Participants) | 217 | 218 | 199
  Grade 3 Rash - Dose 3 | 0 | 0 | 0
  Grade 3 Rash - Across doses | 0 | 0 | 0
  Related Rash - Dose 1: number analyzed (Participants) | 226 | 226 | 207
  Related Rash - Dose 1 | 5 | 6 | 4
  Related Rash - Dose 2: number analyzed (Participants) | 227 | 224 | 207
  Related Rash - Dose 2 | 3 | 2 | 3
  Related Rash - Dose 3: number analyzed (Participants) | 217 | 218 | 199
  Related Rash - Dose 3 | 9 | 4 | 1
  Related Rash - Across doses | 13 | 11 | 7
  Any Urticaria - Dose 1: number analyzed (Participants) | 226 | 226 | 207
  Any Urticaria - Dose 1 | 5 | 3 | 1
  Any Urticaria - Dose 2: number analyzed (Participants) | 227 | 224 | 207
  Any Urticaria - Dose 2 | 2 | 3 | 1
  Any Urticaria - Dose 3: number analyzed (Participants) | 217 | 218 | 199
  Any Urticaria - Dose 3 | 6 | 2 | 1
  Any Urticaria - Across doses | 10 | 7 | 3
  Grade 3 Urticaria - Dose 1: number analyzed (Participants) | 226 | 226 | 207
  Grade 3 Urticaria - Dose 1 | 0 | 0 | 0
  Grade 3 Urticaria - Dose 2: number analyzed (Participants) | 227 | 224 | 207
  Grade 3 Urticaria - Dose 2 | 0 | 0 | 0
  Grade 3 Urticaria - Dose 3: number analyzed (Participants) | 217 | 218 | 199
  Grade 3 Urticaria - Dose 3 | 0 | 0 | 0
  Grade 3 Urticaria - Across doses | 0 | 0 | 0
  Related Urticaria - Dose 1: number analyzed (Participants) | 226 | 226 | 207
  Related Urticaria - Dose 1 | 3 | 1 | 0
  Related Urticaria - Dose 2: number analyzed (Participants) | 227 | 224 | 207
  Related Urticaria - Dose 2 | 2 | 2 | 1
  Related Urticaria - Dose 3: number analyzed (Participants) | 217 | 218 | 199
  Related Urticaria - Dose 3 | 5 | 1 | 1
  Related Urticaria - Across doss | 7 | 4 | 2

7. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 50 millimetres (mm) of injection site.
Time Frame: as for outcome 6
Population: The analysis was based on the TVC, which included all subjects with at least one study vaccine administered, on subjects with symptom sheets completed and for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix (15-25 Years) Group | Cervarix (26-45 Years) Group | Cervarix (46-55 Years) Group
Number analyzed (Participants) | 227 | 226 | 207
Participants
  Any Pain - Dose 1: number analyzed (Participants) | 226 | 226 | 207
  Any Pain - Dose 1 | 197 | 182 | 141
  Any Pain - Dose 2: number analyzed (Participants) | 227 | 224 | 207
  Any Pain - Dose 2 | 186 | 162 | 120
  Any Pain - Dose 3: number analyzed (Participants) | 217 | 218 | 199
  Any Pain - Dose 3 | 179 | 172 | 124
  Any Pain - Across doses | 220 | 210 | 171
  Grade 3 Pain - Dose 1: number analyzed (Participants) | 226 | 226 | 207
  Grade 3 Pain - Dose 1 | 6 | 6 | 3
  Grade 3 Pain - Dose 2: number analyzed (Participants) | 227 | 224 | 207
  Grade 3 Pain - Dose 2 | 11 | 6 | 4
  Grade 3 Pain - Dose 3: number analyzed (Participants) | 217 | 218 | 199
  Grade 3 Pain - Dose 3 | 13 | 7 | 3
  Grade 3 Pain - Across doses | 23 | 15 | 9
  Any Redness - Dose 1: number analyzed (Participants) | 226 | 226 | 207
  Any Redness - Dose 1 | 77 | 80 | 70
  Any Redness - Dose 2: number analyzed (Participants) | 227 | 224 | 207
  Any Redness - Dose 2 | 70 | 80 | 60
  Any Redness - Dose 3: number analyzed (Participants) | 217 | 218 | 199
  Any Redness - Dose 3 | 90 | 85 | 65
  Any Redness - Across doses | 133 | 126 | 101
  Grade 3 Redness - Dose 1: number analyzed (Participants) | 226 | 226 | 207
  Grade 3 Redness - Dose 1 | 0 | 0 | 0
  Grade 3 Redness - Dose 2: number analyzed (Participants) | 227 | 224 | 207
  Grade 3 Redness - Dose 2 | 0 | 4 | 2
  Grade 3 Redness - Dose 3: number analyzed (Participants) | 217 | 218 | 199
  Grade 3 Redness - Dose 3 | 0 | 3 | 0
  Grade 3 Redness - Across doses | 0 | 6 | 2
  Any Swelling - Dose 1: number analyzed (Participants) | 226 | 226 | 207
  Any Swelling - Dose 1 | 36 | 52 | 37
  Any Swelling - Dose 2: number analyzed (Participants) | 227 | 224 | 207
  Any Swelling - Dose 2 | 49 | 61 | 47
  Any Swelling - Dose 3: number analyzed (Participants) | 217 | 218 | 199
  Any Swelling - Dose 3 | 66 | 70 | 60
  Any Swelling - Across doses | 96 | 100 | 83
  Grade 3 Swelling - Dose 1: number analyzed (Participants) | 226 | 226 | 207
  Grade 3 Swelling - Dose 1 | 1 | 0 | 1
  Grade 3 Swelling - Dose 2 | 2 | 3 | 0
  Grade 3 Swelling - Dose 3: number analyzed (Participants) | 217 | 218 | 199
  Grade 3 Swelling - Dose 3 | 0 | 1 | 1
  Grade 3 Swelling - Across doses | 3 | 3 | 1

8. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: During the 30-day (from the day of vaccination up to 29 subsequent days) post-vaccination period
Population: The analysis was based on the TVC, which included all subjects with at least one study vaccine administered and for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix (15-25 Years) Group | Cervarix (26-45 Years) Group | Cervarix (46-55 Years) Group
Number analyzed (Participants) | 229 | 226 | 211
Participants
  Subjects with any AE(s) | 43 | 46 | 28
  Subjects with any Grade 3 AE(s) | 2 | 0 | 4
  Subjects with any Related AE(s) | 13 | 18 | 6

9. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAE)
Description: An SAE is any untoward medical occurrence that resulted in death, was life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity, was a congenital anomaly/birth defect in the offspring of a study subject, or may have evolved into one of the outcomes listed above.
Time Frame: During the entire study period (from Day 0 up to Month 48)
Population: The analysis was based on the TVC (up to Month 7), which included all subjects with at least one study vaccine administered and on the Extended Follow-up (EFU) Vaccinated cohort (Month 7 to Month 48) which included subjects who received 3 doses of vaccine in the primary phase of the study and for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix (15-25 Years) Group | Cervarix (26-45 Years) Group | Cervarix (46-55 Years) Group
Number analyzed (Participants) | 229 | 226 | 211
Participants
  Day 0 to Month 7 | 3 | 1 | 2
  Month 7 to Month 12: number analyzed (Participants) | 213 | 221 | 201
  Month 7 to Month 12 | 0 | 0 | 1
  Month 12 to Month 18: number analyzed (Participants) | 169 | 175 | 180
  Month 12 to Month 18 | 1 | 1 | 4
  Month 18 to Month 24: number analyzed (Participants) | 169 | 181 | 181
  Month 18 to Month 24 | 0 | 1 | 0
  Month 24 to Month 36: number analyzed (Participants) | 162 | 176 | 175
  Month 24 to Month 36 | 3 | 0 | 1
  Month 36 to Month 48: number analyzed (Participants) | 169 | 191 | 181
  Month 36 to Month 48 | 0 | 5 | 5

10. Secondary Outcome: Number of Subjects Reporting New Onset of Chronic Diseases (NOCDs)
Description: NOCDs assessed include chronic diseases such as autoimmune disorders, diabetes, allergies also asthma and pathognomic signs/symptoms of these diseases.
Time Frame: During the entire study period (from Day 0 up to Month 48)
Population: The analysis was based on the TVC (data up to Month 7), which included all subjects with at least one study vaccine administered and on the EFU Vaccinated cohort (data from Month 7 to Month 48) which included subjects who received 3 doses of vaccine in the primary phase of the study and for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix (15-25 Years) Group | Cervarix (26-45 Years) Group | Cervarix (46-55 Years) Group
Number analyzed (Participants) | 229 | 226 | 211
Participants
  Day 0 to Month 7 | 3 | 1 | 0
  Month 7 to Month 12: number analyzed (Participants) | 213 | 221 | 201
  Month 7 to Month 12 | 0 | 0 | 0
  Month 12 to Month 18: number analyzed (Participants) | 169 | 175 | 180
  Month 12 to Month 18 | 1 | 1 | 2
  Month 18 to Month 24: number analyzed (Participants) | 169 | 181 | 181
  Month 18 to Month 24 | 0 | 0 | 0
  Month 24 to Month 36: number analyzed (Participants) | 162 | 176 | 175
  Month 24 to Month 36 | 2 | 2 | 1
  Month 36 to Month 48: number analyzed (Participants) | 169 | 191 | 181
  Month 36 to Month 48 | 1 | 0 | 0

11. Secondary Outcome: Number of Subjects Reporting Medically Significant Conditions
Description: Medically significant conditions are AEs prompting emergency room or physician visits that were not related to common diseases or routine visits for physical examination or vaccination, or SAEs that were not related to common diseases.
Time Frame: During the entire study period (from Day 0 up to Month 48)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix (15-25 Years) Group | Cervarix (26-45 Years) Group | Cervarix (46-55 Years) Group
Number analyzed (Participants) | 229 | 226 | 211
Participants
  Day 0 to Day 29 | 12 | 12 | 11
  Day 30 to Month 7 | 8 | 8 | 10
  Month 7 to Month 12: number analyzed (Participants) | 213 | 221 | 201
  Month 7 to Month 12 | 1 | 3 | 1
  Month 12 to Month 18: number analyzed (Participants) | 169 | 175 | 180
  Month 12 to Month 18 | 3 | 5 | 6
  Month 18 to Month 24: number analyzed (Participants) | 169 | 181 | 181
  Month 18 to Month 24 | 3 | 3 | 2
  Month 24 to Month 36: number analyzed (Participants) | 162 | 176 | 175
  Month 24 to Month 36 | 5 | 4 | 6
  Month 36 to Month 48: number analyzed (Participants) | 169 | 191 | 181
  Month 36 to Month 48 | 1 | 7 | 4

12. Secondary Outcome: Anti-HPV-16/18 Antibody Titers Assessed by ELISA in a Subset of Subjects in Cervical Secretions (CVS) Samples
Description: Anti-HPV 16/18 antibody titers were detected in CVS samples and presented as GMTs, expressed in EL.U/mL based on ELISA.
Time Frame: At Months 18 and 24
Population: The analysis was based on a subset of subjects from the TVC for whom CVS samples were available and who received at least one dose of vaccine in this study.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix (15-25 Years) Group | Cervarix (26-45 Years) Group | Cervarix (46-55 Years) Group
Number analyzed (Participants) | 59 | 51 | 41
EL.U/mL
  Anti-HPV-16 (Month 18): number analyzed (Participants) | 41 | 47 | 39
  Anti-HPV-16 (Month 18) | 63.6 [43.0 to 94.2] | 50.7 [32.7 to 78.5] | 56.1 [36.3 to 86.7]
  Anti-HPV-16 (Month 24) | 59.2 [44.3 to 79.3] | 52.7 [36.5 to 76.2] | 68.8 [41.0 to 115.4]
  Anti-HPV-18 (Month 18): number analyzed (Participants) | 41 | 47 | 39
  Anti-HPV-18 (Month 18) | 28.4 [17.5 to 46.0] | 38.5 [21.5 to 68.9] | 21.2 [15.2 to 29.6]
  Anti-HPV-18 (Month 24) | 23.3 [17.4 to 31.3] | 32.4 [21.5 to 48.8] | 31.2 [19.2 to 50.5]

13. Secondary Outcome: Number of Subjects Seropositive for Total Immunoglobulin-G (IgG) in Blood (Serum) and in Cervical Samples (Secretion) in a Subset of Subjects
Description: Seropositivity was defined as total IgG ≥ 0 microgram per milliliter (µg/mL) and was detected in sera and in CVS samples by ELISA.
Time Frame: At Months 18 and 24
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix (15-25 Years) Group | Cervarix (26-45 Years) Group | Cervarix (46-55 Years) Group
Number analyzed (Participants) | 59 | 51 | 51
Participants
  IgG serum (Month 18): number analyzed (Participants) | 44 | 51 | 51
  IgG serum (Month 18) | 44 | 51 | 51
  IgG serum (Month 24): number analyzed (Participants) | 59 | 51 | 41
  IgG serum (Month 24) | 59 | 51 | 41
  IgG secretion (Month 18): number analyzed (Participants) | 41 | 47 | 39
  IgG secretion (Month 18) | 39 | 47 | 39
  IgG secretion (Month 24): number analyzed (Participants) | 59 | 51 | 41
  IgG secretion (Month 24) | 57 | 50 | 41

14. Secondary Outcome: Number of Subjects Reporting Pregnancies and Outcomes of Reported Pregnancies
Description: Outcomes of pregnancies were: Abnormal infant / Congenital anomaly, Elective termination, Missed abortion, Normal infant, Premature birth, Spontaneous abortion / Miscarriage and Outcome unknown.
Time Frame: During the entire study period (from Day 0 up to Month 48)
Population: The analysis was based on the TVC, which included all subjects with at least one vaccine administration documented and for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix (15-25 Years) Group | Cervarix (26-45 Years) Group | Cervarix (46-55 Years) Group
Number analyzed (Participants) | 229 | 226 | 211
Participants
  Abnormal infant / Congenital anomaly | 0 | 1 | 0
  Elective termination | 0 | 1 | 0
  Missed abortion | 0 | 2 | 0
  Normal infant | 19 | 21 | 1
  Premature birth | 1 | 1 | 0
  Spontaneous abortion / Miscarriage | 1 | 4 | 0
  Outcome unknown | 1 | 1 | 0

ADVERSE EVENTS:
Time Frame: Solicited symptoms: up to Day 7 post vaccination. AEs: up to Day 30 post vaccination. SAEs throughout the study period (up to Month 48).
Description: The number of events for reported SAEs and AEs (all/related) was not available and encoded as equal to the number of subjects affected.
Arm/Group | Cervarix (15-25 Years) Group | Cervarix (26-45 Years) Group | Cervarix (46-55 Years) Group
All-Cause Mortality (participants affected / at risk) | 0/229 | 0/226 | 2/211
Serious Adverse Events (participants affected / at risk) | 6/229 | 8/226 | 11/211
Other Adverse Events (participants affected / at risk) | 224/229 | 216/226 | 182/211
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cervarix (15-25 Years) Group (N=229) | Cervarix (26-45 Years) Group (N=226) | Cervarix (46-55 Years) Group (N=211)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Multiple sclerosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Optic neuritis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Vestibular neuronitis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Carotid artery dissection (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cervical polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Gastroduodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Abortion spontaneous (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 3 (3)
Premature labour (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2) | 0 (0)
Abortion spontaneous complete (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cervarix (15-25 Years) Group (N=229) | Cervarix (26-45 Years) Group (N=226) | Cervarix (46-55 Years) Group (N=211)
Pain (General disorders) | 220 (220) | 210 (210) | 171 (171)
Redness (General disorders) | 133 (133) | 126 (126) | 101 (101)
Swelling (General disorders) | 96 (96) | 100 (100) | 83 (83)
Arthralgia (General disorders) | 45 (45) | 43 (43) | 47 (47)
Fatigue (General disorders) | 128 (128) | 116 (116) | 81 (81)
Fever (General disorders) | 21 (21) | 19 (19) | 5 (5)
Gastrointestinal symptoms (General disorders) | 51 (51) | 33 (33) | 31 (31)
Headache (General disorders) | 123 (123) | 100 (100) | 82 (82)
Myalgia (General disorders) | 126 (126) | 97 (97) | 83 (83)
Rash (General disorders) | 16 (16) | 14 (14) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.